CLINICAL TRIAL: NCT02756676
Title: Impact of an Intensive Multi-Disciplinary Rehabilitation Treatment on Quality Of Life in Subjects With Parkinson's Disease
Brief Title: Impact of Rehabilitation in Quality of Life in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QoL and rehab in PD
Record Dates: First submitted 2016-04-02; First posted 2016-04-29 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Quality of Life; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rehabilitative treatment (MIRT) (Experimental): Rehabilitative treatment MIRT consist in daily sessions of: motor treatment, occupational therapy and language speech therapy
  Interventions: Procedure: Multidisciplinary Intensive Rehabilitation Treatment (MIRT)

INTERVENTIONS:
Procedure: Multidisciplinary Intensive Rehabilitation Treatment (MIRT) — MIRT consists of a 4-week physical therapy that entails four daily sessions, five days a week, in a hospital setting. The duration of each session is about one hour. The first session comprise cardiovascular warm-up activities, relaxation, muscle- stretching, exercises to improve the range of motion of spinal, pelvic and scapular joints, exercises to improve the functionality of the abdominal muscles, and postural changes in the supine position. The second session includes aerobic exercises to improve balance and gait using a stabilometric platform, treadmill plus, crossover and cycloergometer. The third is a session of occupational therapy to improve autonomy in daily living activities. The last session includes one hour of speech therapy.

SUMMARY:
This study is aimed to evaluate the impact of an intensive, multidisciplinary rehabilitative program on quality of life in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive neurodegenerative disease clinically characterized by rigidity, bradykinesia and resting tremor. Beyond these symptoms the principal feature of this condition is the lost of habitual automatic movements and the disruption of different cognitive-motivational processes. These features are related to a pathological dopaminergic tone that alters the cortico-striatal pathways with several consequences on motor and emotional behaviours. Given its complexity PD impact very seriously on patients' quality of life (QoL).

Dopamine replacement therapy (DRT) is the standard treatment for the motor symptom of PD and previous studies have demonstrated its positive effect on QoL. However DRT does not reduce axial PD symptoms such as freezing of gait, postural instability and balance disturbances. Further, long-term DRT could negatively impact on cognitive and motivational functions and leads to different motor and behavioural side effects.

In the last years, rehabilitation has been proposed as an effective and complementary treatment for the management of PD and several evidences highlighted the need of a multidisciplinary and intensive approach to achieve good results.

To evaluate the impact of an intensive, multidisciplinary rehabilitation treatment (MIRT), on QoL of subjects with PD. Literature data showed that this type of treatment determine a positive effect on both motor and non-motor symptoms. Starting from these evidences, in this study the investigators have examined whether MIRT act positively on QoL and for how long this potential positive effect is maintained.

250 PD patients with Parkinson's Disease hospitalized for a 4-weeks MIRT were enrolled. PDQ39 was administered at enrolment, and at three points after discharge: at 1, 3 and 6 months. The investigators decided to evaluate QoL after homecoming in order to avoid an inpatient state bias. Other outcome measures were considered and assessed at the enrolment and at discharge: Unified Parkinson's Disease Scale (UPDRS), Parkinson Disease Disability Scale (PDDS), Berg Balance Scale (BBS), FOG (Freezing of Gait Questionnaire), 6MWT (6 minutes walking Test), Time Up and Go test (TUG). Cognitive and psychopathological status of patients was also assessed using Mini Mental State Examination (MMSE), Frontal Assessment Battery (FAB), State Trait Anxiety Inventory (STAY I-II), Beck Depression Inventory (BDI).

ELIGIBILITY:
Inclusion Criteria:

* Parkinson Disease
* MMSE ≥ 24

Exclusion Criteria:

* Co-morbidity with other neurological disease
* Visual and auditory dysfunctions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Parkinson Disease Questionnaire (PDQ39) | 6 month
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better QoL

SECONDARY OUTCOMES:
Unified Parkinson's disease Rating Scale (UPDRS) | 6 month
six minute walking test (6MWT) | 6 month
Berg Balance Scale (BBS) | 6 month
Freezing of Gait Questionnaire (FoG) | 6 month
Parkinson Disease Disability Scale | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital - Gravedona ed Uniti (CO, Italy)
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gradevole Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrazzoli D, Ortelli P, Zivi I, Cian V, Urso E, Ghilardi MF, Maestri R, Frazzitta G. Efficacy of intensive multidisciplinary rehabilitation in Parkinson's disease: a randomised controlled study. J Neurol Neurosurg Psychiatry. 2018 Aug;89(8):828-835. doi: 10.1136/jnnp-2017-316437. Epub 2018 Jan 10. PMID 29321141